CLINICAL TRIAL: NCT06789406
Title: Post-Market Clinical Follow-up Study of the Axonics SNM System Model 5101 (R20)
Brief Title: PMCF Study of the Axonics SNM System Model 5101 (R20)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Axonics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 105-0104
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Urinary Urge Incontinence (UUI); Urinary Frequency (UF); Overactive Bladder (OAB)
MeSH Terms: conditions — Urinary Incontinence, Urge; Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Overactive Bladder (Other): Participants with the Axonics SNM System Model 5101 and followed up regarding their overactive bladder symptoms.
  Interventions: Device: Axonics SNM System INS Model 5101 (R20)

INTERVENTIONS:
Device: Axonics SNM System INS Model 5101 (R20) — Participants treated with the rechargeable Axonics SNM System Model 5101 also referred to as R20. Commercial devices used in this study are within their intended use as described in each geography's approved instructions for use.

SUMMARY:
Post-market clinical follow-up for continued assessment of safety and performance to confirm long-term outcomes of the Axonics SNM System INS Model 5101.

DETAILED DESCRIPTION:
This post-market clinical follow-up (PMCF) is conducted to assess the continued safety, device performance, and clinical benefit of the rechargeable Axonics SNM System INS Model 5101 also referred to as R20.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older
2. Primary indication of OAB (urinary urgency incontinence (UUI) / urinary frequency (UF) who are not candidates for, or who have failed conservative treatment
3. Willing and capable to provide written consent and agrees to comply with specified evaluations at clinical centers for all follow-up assessments

Exclusion Criteria:

1. Any significant medical condition that is likely to interfere with procedures, device operation, or likely to confound evaluation of endpoints (i.e., neurological conditions such as multiple sclerosis)
2. Any psychiatric or personality disorder that is likely to interfere with procedures at the discretion of the participating physician; this may include poor understanding or compliance with requirements
3. Previously underwent an external sacral neuromodulation SNM trial and was deemed a non-responder or was previously implanted with a sacral neuromodulation device and did not get therapeutic benefit (a non-responder)
4. History of allergic response to titanium, zirconia, polyurethane, epoxy, or silicone
5. A female who is breastfeeding
6. A female with a positive urine pregnancy test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2025-09-18 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2031-10 (Estimated)

PRIMARY OUTCOMES:
Performance/Effectiveness - Improvement in Qualify of Life scoring (OAB) | 3 months
  To demonstrate an improvement in Overactive Bladder Quality of Life using the International Consultation of Incontinence Questionnaire Overactive Bladder Qualify of Life (ICIQ-OABqol): questions in each subscale are scored by a summed range of 0 to 100, with a higher score indicating better quality of life. Overall score ≥ 10 points from baseline to follow-up is indicative of a clinically meaningful improvement.
Adverse event reporting (Safety) | 3 months
  Device related, procedure-related and all serious adverse events

SECONDARY OUTCOMES:
Performance/Effectiveness - Improvement in Qualify of Life scoring (OAB) | 12 months
  To demonstrate an improvement in Overactive Bladder Quality of Life using the International Consultation of Incontinence Questionnaire Overactive Bladder Qualify of Life (ICIQ-OABqol): questions in each subscale are scored by a summed range of 0 to 100, with a higher score indicating better quality of life. Overall score ≥ 10 points from baseline to follow-up is indicative of a clinically meaningful improvement.
Performance/Effectiveness - Improvement in Qualify of Life scoring (FI) | 12 months
  Cleveland Clinic Florida - Fecal Incontinence Score (CCF-FIS): scores range from 0 for full continence to 20 for complete incontinence. A higher score is indicative of the severity of fecal incontinence. Assessed if participant had a score of ≥6 at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Mahreen Pakzad, MD, Principal Investigator — University College London Hospitals; Gita Ghadimi, OD, Study Director — Boston Scientific Corporation
Locations (4):
- University of Chicago, Chicago, Illinois, United States
- United Kingdom (3):
  - Bradford Royal Infirmary, Bradford, West Yorkshire
  - Pinderfields Hospital, Wakefield, West Yorkshire
  - University College London Hospital, London

IPD SHARING:
Plan to Share IPD: No